CLINICAL TRIAL: NCT06816017
Title: A Phase I/II, Open-label, Dose Escalation and Extension Study of Intravesical Eciskafusp Alfa in Combination With Bacillus Calmette-guerin (BCG) in Participants With BCG-unresponsive High-risk Non-muscle Invasive Bladder Cancer (NMIBC)
Brief Title: A Study to Evaluate Eciskafusp Alfa in Combination With Bacillus Calmette-guerin (BCG) in Participants With BCG-unresponsive High-risk Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision of the Sponsor.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP45381; 2024-515410-41-00 (Other: EU Trial Number)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-06-16 (Actual); Status verified 2025-06

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: BCG-unresponsive Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I: Dose Escalation (Experimental): Participants will receive multiple ascending doses of eciskafusp alfa in combination with a fixed dose of BCG administered as an intravesicular instillation up to a maximum of 25 months or until detection of high-risk disease or disease progression, toxicity, or withdrawal from study treatment for other reasons, whichever occurs first.
  Interventions: Drug: Eciskafusp Alfa; Drug: BCG Medac Strain
- Phase II: Dose Extension (Cohort A) (Experimental): Participants will receive eciskafusp alfa at the maximum tolerated dose (MTD) and/or the recommended dose for extension (RDE), as determined in Phase 1, in combination with a fixed dose of BCG administered as an intravesical instillation up to a maximum of 25 months or until detection of high-risk disease or disease progression, toxicity, or withdrawal from study treatment for other reasons, whichever occurs first.
  Interventions: Drug: Eciskafusp Alfa; Drug: BCG Medac Strain
- Phase II: Dose Extension (Cohort B) (Experimental): Participants will receive eciskafusp alfa as monotherapy at the MTD or RDE determined in Phase 1, administered as an intravesical instillation up to a maximum of 25 months or until detection of high-risk disease or disease progression, toxicity, or withdrawal from study treatment for other reasons, whichever occurs first.
  Interventions: Drug: Eciskafusp Alfa

INTERVENTIONS:
Drug: Eciskafusp Alfa — Participants will receive eciskafusp alfa via intravesical instillation.
  Other Names: RO7284755
Drug: BCG Medac Strain — Participants will receive BCG via intravesical instillation.
  Arms: Phase I: Dose Escalation; Phase II: Dose Extension (Cohort A)

SUMMARY:
The study aims to establish the safety, tolerability, pharmacokinetics (PK), relevant biomarkers, pharmacodynamics (PD) and preliminary anti-tumor activity of the intravesical administration of eciskafusp alfa in combination with BCG in participants with BCG-unresponsive high-risk NMIBC.

The study plans a similar evaluation of eciskafusp alfa in monotherapy following a positive interim analysis of the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed high risk non muscle invasive transitional cell carcinoma classified according to World Health Organization (WHO) grading system
* Absence of resectable disease after transurethral resection of bladder tumor (TURBT) procedures
* The most recent cystoscopy/TURBT must have been performed within 12 weeks and up to 14 days of the first dose of study treatment
* Presence of BCG-unresponsive disease defined as persistent or recurrent carcinoma in situ [CIS] (± recurrent Ta/T1 disease) within 12 months of receiving adequate BCG therapy
* The participant is considered ineligible for radical cystectomy or has elected not to undergo the procedure.
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb) test at screening
* Negative hepatitis C virus (HCV) antibody test at screening

Exclusion Criteria:

* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Active infections (both systemic and local urinary)
* Congenital or acquired immune deficiencies resulting in immunosuppression
* Known human immunodeficiency virus (HIV) infection
* History of radiotherapy of the bladder
* History of perforation of the bladder
* Major surgery or significant traumatic injury within 28 days prior to first administration of study treatment or anticipation of the need for major surgery during treatment
* Participants currently receiving investigational or commercial anti-cancer agents or anti-cancer therapies other than BCG, and supportive care therapies for active disease
* Any intervening intravesical immunotherapy or chemotherapy from the time of the most recent cytoscopy/TURBT to the start of study treatment
* Systemic immune-modulating and systemic immunosuppressive agents/medication
* Administration of a live, attenuated vaccine within 28 days prior to first administration of study treatment
* Recurrence of BCG unresponsive CIS > 12 months after last BCG instillation
* Concurrent second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Number of Participants With Adverse Events (AEs) | From Baseline (Day 1) up to 28 days after final dose of study treatment (up to Month 26)
Phase I: Number of Participants With Dose Limiting Toxicities (DLTs) | From Day 1 up to Day 14
Phase I: Recommended Dose for Extension (RDE) of Eciskafusp Alfa in Combination With BCG | At Month 25
Phase II (Cohort A): Complete Response Rate (CRR) at 12 Months | At Month 12

SECONDARY OUTCOMES:
Phase I and Phase II: CRR at any Time | Up to Month 36
Phase I and Phase II: CRR at 6, 18 and 24 Months | At Months 6, 18 and 24
Phase I and Phase II (Cohort B): CRR at 12 Months | At Month 12
Phase I and Phase II: Duration of Response (DOR) | Time from the first occurrence of a documented CR until the time of evidence that the participant no longer meets the definition for CR or death from any cause, whichever occurs first (up to Month 36)
Phase I and Phase II: DOR Rate at Specific Timepoints | At Months 6, 12, 18, 24, 30 and 36
Phase I and Phase II: Time to Worsening of NMIBC Grade or Stage, or Death | Time from the first dose of study treatment to the first occurrence of documented worsening of grade, stage or death from any cause, whichever occurs first (up to Month 36)
Phase I and Phase II: Progression Free Survival (PFS) to Muscle Invasive or Metastatic Disease or Death | Time from the first dose of study treatment to the first occurrence of documented muscle-invasive or metastatic disease or death from any cause, whichever occurs first (up to Month 36)
Phase I and II: Time to Cystectomy | Time from the first dose of study treatment to the first occurrence of documented cystectomy or death from any cause, whichever occurs first (up to Month 36)
Phase II: Number of Participants With AEs | From Baseline (Day 1) up to 28 days after final dose of study treatment (up to Month 26)
Phase I and Phase II: Number of Participants With Anti-drug Antibodies (ADAs) to Eciskafusp Alfa | Up to Month 36
Phase II: Programmed Cell Death Ligand 1 (PD-L1) Expression in the Tumor Microenvironment (TME) Pre-treatment and During the Study | Predose (-12 weeks to -14 days or archival) and Postdose at Month 6
  PD-L1 expression may be assessed at other timepoints when on-treatment biopsies will be collected.
Phase II: Number of Participants With Cluster of Differentiation 8+ (CD8+) T cell in TME | Predose (-12 weeks to -14 days or archival)
Phase II: Baseline Urine Tumor Deoxyribonucleic Acid (DNA) | Baseline (Day 1 predose)
Phase II: Amount of Urine Tumor DNA at Baseline and During the Study | Up to Month 25

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Macquarie University Hospital, Macquarie Park, New South Wales, Australia
- A.O.U di Verona Policlinico G.B. Rossi, Verona, Veneto, Italy
- Hospital Umum Sarawak, Kuching, Sarawak, Malaysia
- Netherlands (2):
  - NKI/AvL, Amsterdam
  - UMC St Radboud, Nijmegen
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - AIDPORT Sp. z o. o., Skórzewo
- Spain (2):
  - Hospital Univ. 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing.